CLINICAL TRIAL: NCT02054663
Title: Transition From Ticagrelor to Clopidogrel Following Acute Coronary Syndrome: To Bolus or Not? The CAPITAL OPTI-CROSS Study.
Brief Title: Transition From Ticagrelor to Clopidogrel Following Acute Coronary Syndrome: To Bolus or Not?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Derek So, Associate Professor, Staff Interventional cardiologist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130605-01H
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Coronary artery disease; Antiplatelet therapy; Ticagrelor; Clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bolus (Experimental): Patients randomized to this arm will receive a 600mg bolus dose of clopidogrel at the time of switching from ticagrelor to clopidogrel, followed by 75mg daily.
  Interventions: Drug: Clopidogrel
- no bolus (Experimental): Individuals randomized to this arm will receive 75mg of clopidogrel at the time of the transition followed by a daily dose of 75mg orally.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Patients on ticagrelor following an acute coronary syndrome, being transitioned to clopidogrel will be randomized to either a one time 600mg bolous dose of clopidogrel followed by 75mg daily or just starting at 75mg daily without a bolous dose.
  Other Names: Plavix

SUMMARY:
After a heart attack patients are routinely started on drugs to inhibit platelets. Ticagrelor is a powerful anti-platelet drug with clinical benefits. However it must be discontinued in some, because of increased risk of bleeding or intolerance. These patients need to be transitioned to another agent, such as Clopidogrel. At present, there is no clinical consensus on the optimal strategy for this switch. Some clinicians elect to give a bolus dose of clopidogrel with 600mg, while others start directly with a 75mg daily dose, with no evidence regarding the benefits or potential complications associated with each strategy. The present proposal will evaluate the pharmacodynamics of 2 strategies with specialized platelet function testing. We hypothesize that a bolus dose of clopidogrel during the switch will confer better ischemic protection without increasing bleeding risk for patients undergoing a switch in therapy.

DETAILED DESCRIPTION:
The overall objective is to evaluate the need for a clopidogrel bolus dose among patients being switched from a regimen of ticagrelor to clopidogrel. In a randomized pharmacodynamics study of 48 patients, we will conduct serial measurements of platelet function/inhibition using the Accumetrics Verifynow assay (platelet inhibition will be expressed as P2Y12 reaction unit [PRU]). Platelet inhibition will be assessed at specific time points over the first 72 hours following the change in medications, which will enable us to determine whether patients in the 2 different strategies may be at increased ischemic or bleeding risks. We hypothesize that a bolus dose of clopidogrel during the switch will confer better ischemic protection without increasing bleeding risk for patients undergoing a switch in therapy.

SPECIFIC AIMS:

1. Primary Aim: To determine with platelet function testing the pharmacodynamics effects of a 600mg bolus dose of clopidogrel compared with no bolusing among patients being switched from ticagrelor to clopidogrel.
2. To determine if patients receiving a clopidogrel bolus have improvement in ischemic protection relative to patients without a bolus dose.
3. To determine if patients receiving a clopidogrel bolus may be exposed to increase bleeding risk relative to those without a bolus dose.

ELIGIBILITY:
Inclusion Criteria:

* age > 18,
* admission for acute coronary syndrome,
* on dual anti-platelet therapy (including ticagrelor)
* Being transitioned to clopidogrel by their treating physician
* provided informed consent

Exclusion Criteria:

* Bleeding/intolerance to clopidogrel
* Thrombocytopenia (platelet count < 100, 000 per uL)
* Hematocrit <30% or >52%
* treatment with glycoprotein IIb/IIIa inhibitor, 24 hours prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition as assessed by P2Y12 reaction Unit (PRU) after transition from Ticagrelor to Clopidogrel. | 72 hours
  Post randomization, blood samples at scheduled time points will be collected. Samples would enable measurement of platelet inhibition using the VerifyNow P2Y12 assay. Blood samples will be collected at baseline (prior to clopidogrel dose), 12, 24, 48, 54, 60 and 72 hours post initiation of therapy. The primary endpoint is the difference in platelet inhibition between our 2 different groups (bolus vs no bolus), as measured by P2Y12 reaction unit (PRU) using the VerifyNow assay. The PRUs have now been widely used and accepted as a measure of platelet function in the research setting. PRU will be collected at the above mentioned time points. The primary outcome will be platelet function expressed as PRUs as a continuous variable over the 72 hour time period and compared between the 2 groups.

SECONDARY OUTCOMES:
The difference in platelet inhibition (as expresses as PRU) between the two groups at specified time points. | 72 hours
  In the secondary outcome mean platelet inhibition as measured by PRU will be compared at each specified time point between the the 2 groups.

OTHER OUTCOMES:
Differences in clinical outcomes between the 2 groups within 30 days post transition. | 30 days post transition
  Other secondary clinical endpoints include the following.
  1. TIMI major bleed
  2. TIMI minor bleed
  3. Myocardial Infarction
  4. Stroke
  5. Stent thrombosis
  6. Death
  patients will be contacted on day 30 via telephone and asked about any bleeding complications, need for transfusions, recurrent chest pains, hospitalizations or treatment as acute coronary syndrome (including repeat angiography). New onset neurological symptoms in keeping acute cerebral accidents or hospitalization for a cerebral accident.

CONTACTS AND LOCATIONS:
Overall Officials: Derek So, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Pourdjabbar A, Hibbert B, Chong AY, Le May MR, Labinaz M, Simard T, Ramirez FD, Lugomirski P, Maze R, Froeschl M, Glover C, Dick A, Marquis JF, Bernick J, Wells G, So DY; CAPITAL Investigators. A randomised study for optimising crossover from ticagrelor to clopidogrel in patients with acute coronary syndrome. The CAPITAL OPTI-CROSS Study. Thromb Haemost. 2017 Jan 26;117(2):303-310. doi: 10.1160/TH16-04-0340. Epub 2016 Oct 20. PMID 27761582